CLINICAL TRIAL: NCT02134704
Title: Kinematic Analysis of the Trunk in Patients With Moderate Scoliosis
Brief Title: MOUVSCO: Kinematic Analysis of the Trunk in Patients With Moderate Scoliosis
Acronym: MOUVSCO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All patients were recruted but it has been difficulte to recrute all volunteers (15/30) . However data should be sufficient for analyse of data.
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other); Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MOUVSCO-DCIC-1411
Record Dates: First submitted 2014-05-05; First posted 2014-05-09 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scoliosis Group (Experimental)
  Interventions: Other: Data recording with all sensors
- Healthy Volunteers Group (Experimental)
  Interventions: Other: Data recording with all sensors

INTERVENTIONS:
Other: Data recording with all sensors — The sensors will be placed in the child body and will allow the collection of all the data of the trial.

SUMMARY:
The hypothesis of this study is that moderate scoliosis patients have postural and kinematic differences (static and dynamic) compared with healthy volunteers and it is possible to characterize and quantify.

The aim of this study is the detailed analysis of postural anomalies in moderate scoliosis patients compared with healthy volunteers

DETAILED DESCRIPTION:
Subjects participating in the study must wear sensors that will be arrange at the shoulders, spine, pelvis and legs. Subjects will perform under the direction of the investigator, different tasks of a total duration of 45 minutes.

During the period of experimentation, the data collected will be:

* the positions of each one of the sensors in all three planes of space,
* the ground support forces

ELIGIBILITY:
Scoliosis Group - Inclusion Criteria:

* female children patients from 9 to 16 years old,
* patients with idiopathic scoliosis lumbar left and / or right thoracic,
* patients with moderate scoliosis: Cobb angle measured on a radiograph between 10 ° and 25°,
* both parents of patients must be affiliated to social security or similarly regime.

Healthy Volunteers Group - Inclusion Criteria:

* female children from 9 to 16 years old, matched in age and size with scoliosis patients,
* children with no neuromuscular disease that may have an influence on the required tasks,
* both parents of children must be affiliated to social security or similarly regime,

Exclusion Criteria:

* refusal to consent: from child's in age to consent or from both parents

Ages: 9 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Relative movements, in mm, of the spinous processes in the three planes of space | 2 hours
  Characterize the kinematic anomalies in scoliosis patients compared with healthy volunteers during typical tasks of trunk flexion.

SECONDARY OUTCOMES:
Relative rotations of the bi-acromial line, thoracic and pelvic plan. | 2 hours
  * Assess the existence of kinematic differences between the scoliosis patients and healthy volunteers during forward bending.
  * Assess the kinematic differences between the scoliosis patients and healthy volunteers when they sit and up from a stool.
  * Assess the kinematic differences between the scoliosis patients and healthy volunteers during walking.
Walking speed, step length and single stance time. | 2 hours
  Assess the performance of walking in scoliosis patients.
The surface of displacement of the center of plantar pressure, static relative orientation of the bi-acromial line, thoracic and pelvic plan. | 2 hours
  Assess balance and static posture of scoliotic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelien Courvoisier, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Émilie Chipon, Grenoble, Isère, France

REFERENCES:
- See also: Website of the Grenoble clinical investigation center - Technological Innovation — http://www.cic-it-grenoble.fr/